CLINICAL TRIAL: NCT06791005
Title: A Comparative Study of Preoperative and Intraoperative Carbon Nanoparticles Injection in Patients Undergoing Thyroid Cancer Surgery
Brief Title: A Clinical Study on the Benefits of Carbon Nanoparticles Injection Time in Patients With Thyroid Cancer.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: nanoc
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Papillary Thyroid Cancer
Keywords: Papillary Thyroid Cancer; thyroid surgery; developer; complication
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Preoperative Injection Before Partial Thyroidectomy Group (Experimental): Patients in this group will undergo partial thyroidectomy and preoperative injection of carbon nanoparticles.
  Interventions: Drug: Preoperative Injection of Carbon Nanoparticles
- Intraoperative Injection During Partial Thyroidectomy Group (Active Comparator): Patients in this group will undergo partial thyroidectomy and intraoperative injection of carbon nanoparticles.
  Interventions: Drug: Intraoperative Injection of Carbon Nanoparticles
- Preoperative Injection Before Total Thyroidectomy Group (Experimental): Patients in this group will undergo total thyroidectomy and preoperative injection of carbon nanoparticles.
  Interventions: Drug: Preoperative Injection of Carbon Nanoparticles
- Intraoperative Injection During Total Thyroidectomy Group (Active Comparator): Patients in this group will undergo total thyroidectomy and intraoperative injection of carbon nanoparticles.
  Interventions: Drug: Intraoperative Injection of Carbon Nanoparticles

INTERVENTIONS:
Drug: Preoperative Injection of Carbon Nanoparticles — 1.Medication: Carbon nanoparticles, Chongqing Lemay Pharmaceutical Co. Ltd., production license, Food and Drug Administration Production License No. (China) 2007204, Registration No.: State prescription H20041829. The product is a stable suspension of carbon particles with a diameter of 150 nm.2. 2.Preoperative injection method: The preoperative subgroup was injected with carbon nanoparticles 2-6 hours before surgery, with the patient in the position of padded shoulder, and disinfection around the puncture point was prepared prior to the injection of carbon nanoparticles. Under ultrasound guidance, a fine needle was used to puncture the lower 1/3 of the ventral surface, and no blood was detected on aspiration, i.e., 0.1 mL of carbon nanoparticles was injected into each of the 2 sites of each gland, and the total volume of carbon nanoparticles injected was 0.4 mL, and the depth of injection was approximately within the upper third of the gland.
  Arms: Preoperative Injection Before Partial Thyroidectomy Group; Preoperative Injection Before Total Thyroidectomy Group
Drug: Intraoperative Injection of Carbon Nanoparticles — Intraoperative injection of carbon nanoparticles: After exposing the thyroid peritoneum, 0.1 mL of carbon nanoparticles was injected into both sides of normal thyroid tissue using a syringe (1 mL). Two spots were needed for each flap, and the total volume of injected carbon nanoparticles was 0.4 mL. Finally, the needle was gently backed up under negative pressure to prevent the leakage of carbon nanoparticles.
  Arms: Intraoperative Injection During Partial Thyroidectomy Group; Intraoperative Injection During Total Thyroidectomy Group

SUMMARY:
The detection rate of thyroid cancer (PTC) has increased rapidly in recent years. Except undifferentiated cancer, surgery is still one of the most important treatments for all types of thyroid cancer, and there is a consensus to use the lobes of the gland as the minimum extent of resection. In the meantime, a basic consensus has been reached that central zone lymph node (VI) dissection is the minimum extent of lymph node dissection. In clinical practice, neck surgery and lumpectomy are mostly performed. Hypoparathyroidism and recurrent laryngeal nerve injury are the most common complications of radical surgery for thyroid cancer, both in open surgery and the luminal approach. Once these complications occur, they have a serious impact on the quality of life of patients in the postoperative period. A number of contrast agents are now being used to help minimize complications. Carbon nanoparticles are an effective and non-harmful negative developer, and many studies have confirmed that carbon nanoparticles can be used to identify parathyroid glands in thyroid surgery. Intraoperative injection of nanocarbon is effective in increasing the quality of intraoperative parathyroid detection and lymph node clearance and reducing adverse effects, such as postoperative hypokalemia.However, there is no complete clinical guideline for preoperative intraglandular injection of carbon nanoparticles, and there is no standardized dosage for appropriate injection time, injection dose, and injection method. At the same time, there is still the problem of carbon nanoparticle leakage. At our medical center, we have found that preoperative injection of carbon nanoparticles via ultrasound-guided fine needle puncture may yield better results by reducing CNS exudation in the surgical area. In this study, we will collect more than 400 patients who underwent thyroidectomy in 2025 and underwent carbon nanoparticle injections at different time points and analyzed their intraoperative and postoperative conditions as a basis for analyzing the difference in patient benefits between preoperative and intraoperative carbon nanoparticle injections and to provide data to support the clinical use of carbon nanoparticles.

DETAILED DESCRIPTION:
1. Use of drugs: Carbon nanoparticles, Chongqing Lemay Pharmaceutical Co. Ltd., production license, Food and Drug Administration Production License No. (China) 2007204, Registration No.: State prescription H20041829. The product is a stable suspension of carbon particles with a diameter of 150 nm.2. Preoperative injection method: The preoperative subgroup was injected with carbon nanoparticles 2-6 hours before surgery, with the patient in the position of padded shoulder, and disinfection around the puncture point was prepared prior to the injection of carbon nanoparticles. Under ultrasound guidance, a fine needle was used to puncture the lower 1/3 of the ventral surface, and no blood was detected on aspiration, i.e., 0.1 mL of carbon nanoparticles was injected into each of the 2 sites of each gland, and the total volume of carbon nanoparticles injected was 0.4 mL, and the depth of injection was approximately within the upper third of the gland.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative pathological assessment indicated the presence of thyroid cancer with a maximum diameter of less than 4 cm.
* Postoperative pathological evaluation confirmed bilateral thyroid cancer or lateral lymph node metastasis.
* Vocal cord examination conducted one week prior to surgery revealed no abnormalities.
* The patient had no history of prior thyroid surgery and required a total thyroidectomy.
* Blood pressure was stably controlled.
* The patient regained consciousness and was able to communicate normally.

Exclusion Criteria:

* Prior to enrollment, the patient had received radiotherapy, chemotherapy, or isotope therapy.
* A documented history of thyroid surgery.
* Age under 16 years.
* Known allergies to the medications under investigation or an inability to tolerate surgical intervention.
* Presence of a retrosternal thyroid tumor.
* Tumor invasion of the parathyroid glands and/or the recurrent laryngeal nerve during surgical procedures.
* Postoperative pathology suggestive of medullary carcinoma or undifferentiated carcinoma.
* Development of a postoperative tracheal fistula.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
age | up to three years
  Age will be aggregated using "years" as the unit of measurement.
Genders | up to three years
  Data will be summarized in terms of "male" and "female" as units of measurement.
Height | up to three years
  The height indicator will summarize the data in "meters".
Weight | up to three years
  The weight indicator will summarize data in "kilograms".
BMI | up to three years
  BMI will be summarized in "kg/m^2".
Tumor Diameter Size | up to three years
  Tumor diameter size will be summarized in "millimeters".
Tumor Location | up to three years
  Data will be summarized in terms of "Upper pole of left lobe" , "middle pole of left lobe" , "lower pole of left lobe" , "upper pole of right lobe" , "middle pole of right lobe" , "lower pole of right lobe" , "isthmus" and "multifocal" as units of measurement.
Pathological Results | up to three years
  Data will be summarized in terms of detailed pathological results and "none" .
Preoperative Serum Calcium | up to three years
  The Calcium indicator will summarize data in "mmol/L".
Preoperative Serum Thyroid Hormone | up to three years
  The thyroid hormone indicator will summarize data in "pmol/L".
Preoperative Serum Parathyroid Hormone | up to three years
  The parathyroid hormone will summarize data in "pmol/L".
Preoperative serum TSH | up to three years
  The TSH indicator will summarize data in "mlU/L".
Preoperative Vocal Cord Movement Problems or Laryngoscopy Result | up to three years
  Data will be summarized in terms of "normal" , "symptomatic" and "laryngoscopy abnormal" as units of measurement.
Carbon Nanoparticles Injection Site | up to three years
  Data will be summarized in terms of "Upper pole of left lobe" , "middle pole of left lobe" , "lower pole of left lobe" , "upper pole of right lobe" , "middle pole of right lobe" , "lower pole of right lobe" , "isthmus" and "multi-site injection" as units of measurement.
Number of Carbon Nanoparticles Injections | up to three years
  Number of Carbon Nanoparticles Injections
Carbon Nanoparticles Injection Dose | up to three years
  Injection dose will be summarized in "milliliter".
Duration of The Operation | up to three years
  The duration of the operation will summarize data in "h". The time interval from the induction of anesthesia to the end of surgery was selected as the length of surgery, according to the surgical care records
Number of Lymph Node Dissection | up to three years
  Record the total number of lymph nodes dissected, the number of lymph nodes dissected in the central region, the number of lymph nodes dissected in the lateral cervical region and the number of metastatic lymph nodes detected.
Intraoperative Hemorrhage | up to three years
  The intraoperative hemorrhage will summarize data in "milliliter".
Thyroid Staining | up to three years
  Data will be summarized in terms of "A" ,"B" and "C" as units of measurement. A.The stained thyroid is good in the center and at the margins, with clear staining at the edges; B.The stained thyroid gland has good central staining, and the margins are grossly stained, so that the marginal pattern can be roughly observed; C.The stained thyroid stains well, with poorly stained margins;
Lymph node staining | up to three years
  Data will be summarized in terms of "A" ,"B" and "C" as units of measurement. A.The center and margins of the stained lymph nodes are well stained, and the margins are clearly stained; B. The stained lymph nodes have good central staining and grossly stained margins; the marginal pattern can be roughly observed, and the lymph nodes are definite on palpation; C.Good central staining of the stained lymph nodes, unclear staining of the margins, and precise palpation of the lymph nodes.
Parathyroid Glands Staining | up to three years
  Data will be summarized in terms of "A" ,"B" and "C" as units of measurement. A.Good central infiltration, uniform and clear staining throughout the gland; B.Central infiltration is good, staining of the entire gland is still uniform, but flaky stained areas are seen, and the gland is exact on palpation; C.Central infiltration is fair, staining of the entire gland is stellate with no obvious shape, and the gland is exact on palpation.
Nanocarbon Leakage | up to three years
  Data will be summarized in terms of "A" ,"B" and "C" as units of measurement. A.no visible leakage, only slight leakage at the injection site, not affecting the parathyroid glands or the recurrent laryngeal nerve; B.leakage is present and visible to the naked eye, but less than 1/2 of the entire operative field, with staining of the trachea, thyroid peritoneum, and anterior cervical musculature; C.Leakage is present and reaches 1/2 of the entire operative field or Carbon Nanoparticles results in staining of the parathyroid glands or the recurrent laryngeal nerve, affecting identification.
Duration of Postoperative Pain | up to three years
  The duration of postoperative pain will summarize data in "days".
Postoperative Drainage | up to three years
  The postoperative drainage will summarize data in "milliliter".
Length of Postoperative Hospitalization | up to three years
  The length of postoperative hospitalization will summarize data in "days"
Postoperative Serum Parathyroid Hormone | up to three years
  The parathyroid hormone will summarize data in "pmol/L".
Numbness of The Hands and Feet | up to three years
  The numbness of the hands and feet will be summarized with a "yes" or "no" to the data.
Postoperative Laryngeal Recurrent Nerve Irritation and Injury | up to three years
  Postoperative laryngeal recurrent nerve irritation and injury will be summarized with a "yes" or "no" to the data.
Postoperative Hematoma | up to three years
  The postoperative hematoma will be summarized with a "yes" or "no" to the data.
Postoperative Tracheocutaneous Fistula | up to three years
  The postoperative tracheocutaneous fistula will be summarized with a "yes" or "no" to the data.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

DOCUMENTS (2):
  • Study Protocol (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT06791005/Prot_000.pdf
  • Informed Consent Form (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT06791005/ICF_001.pdf